CLINICAL TRIAL: NCT02649400
Title: Assessment of Functional Capacity, Inflammatory Markers and Autonomic Function in Women With Heart Failure With Preserved Ejection Fraction and Previous Coronary Artery Disease
Brief Title: Assessment of Functional Capacity and Inflammatory Markers in Women With Heart Failure With Preserved Ejection Fraction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Daniel Figueiredo Alves da Silva, Post-graduate Student, Federal University of São Paulo
Other Study IDs: 15218913.6.0000.5505
Record Dates: First submitted 2015-12-02; First posted 2016-01-07 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure, Diastolic; Coronary Artery Disease; Inflammation
MeSH Terms: conditions — Heart Failure, Diastolic; Coronary Artery Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood and plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diastolic Heart Failure: Women with diastolic heart failure and previous coronary artery disease

SUMMARY:
This study assesses the impact of diastolic heart failure on exercise capacity in women who have a previous coronary condition. All the participants will go through the same evaluation.

DETAILED DESCRIPTION:
It is well established that systolic heart failure impacts exercise capacity and quality of life, diastolic heart failure however, is not well documented as a condition that reduces physical performance.

To confirm that patients have a diastolic disfunction an echocardiography will be performed, this will also yield the left ventricle ejection fraction to confirm the preserved ejection fraction heart failure diagnostics.

Exercise capacity will be assessed using the distance walked on the six-minute walking test, performed on a 30m corridor.

Pulmonary function will be assessed with spirometry and values of forced vital capacity and forced expired volume in one second will be recorded and compared to the age-predicted values.

Respiratory strength will be determined by maximal pressure achieved on a respiratory manometer.

Peripheral muscular strength will be assessed with a handheld dynamometer. Knee extension strength of the dominant leg will be recorded.

An echocardiography will be performed to assess systolic and diastolic function and ejection fraction.

Heart autonomic function will be evaluated using a heart rate monitor and a computer software to identify the sympathovagal balance.

ELIGIBILITY:
Inclusion Criteria:

* Women;
* Aged between 35 and 70 years;
* Coronary artery disease proven by coronary angiography;
* Diastolic heart failure confirmed by recent echocardiography (6 months);
* Left Ventricle ejection fraction of greater than 50%;
* Absence of acute or chronic pulmonary disease;
* Patient clinically compensated;
* Consent form signed for participation in the research

Exclusion Criteria:

* Inability to perform spirometry;
* Presence of acute or chronic pulmonary disease;
* Chronic inflammatory disease, kidney or liver disease;
* Patients using corticosteroids, aspirin or other nonsteroidal anti-inflammatory;
* Clinical or laboratory evidence of infection;
* Morbid obesity;
* Hemodynamic instability at the time of spirometry;
* Patient's or legal guardian request to leave at any time of the study.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with coronary artery disease diagnosed through angiography and heart failure with preserved ejection fraction diagnosed via ecocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | Up to 1 year after diagnosis
  Measured by the distance walked in the six-minute walking test in meters.
Inflammatory markers | Up to 1 year after diagnosis on the same day as functional capacity assessment
  Inflammatory markers evaluated using specific assays for blood analysis Interleukin (IL) 1 (pg/mL), IL-6 (pg/mL), IL 8 (pg/mL),Tumor Necrosis Factor alpha (pg/mL), Brain Natriuretic Peptide (BNP) (pg/mL), pro-BNP (pg/mL);
  Lab results will be analysed for each marker and values will be compared to laboratory reference data to identify values out of range.
Inflammatory Markers | Up to 1 year after diagnosis on the same day as functional capacity assessment
  Inflammatory markers evaluated using specific assays for blood analysis for high sensitivity C reactive protein (mg/L), alpha-1-acid glycoprotein (mg/dL) and platelets (platelets/cubic millimeters), lactate (mg/dL), uric acid (mg/dL)

SECONDARY OUTCOMES:
Heart autonomic function | Up to 1 year after diagnosis on the same day as functional capacity assessment
  Sympathovagal balance assessed by heart rate variability using a heart monitor
Quality of life | Up to 1 year after diagnosis on the same day as functional capacity assessment
  Quality of life assessed by the Minnesota questionnaire specific for heart failure
Pulmonary function | Up to 1 year after diagnosis on the same day as functional capacity assessment
  Pulmonary function assessed by spirometry for obtaining values of forced expired volume in one second (FEV1), forced vital capacity (FVC) and FEV1/FVC ratio
Respiratory muscle strength | Up to 1 year after diagnosis on the same day as functional capacity assessment
  Respiratory muscle strength assessed by manometer for obtaining maximal inspiratory pressure and maximal expiratory pressure values in cmH2O.
Peripheral muscle strength | Up to 1 year after diagnosis on the same day as functional capacity assessment
  Peripheral muscle strength assessed by the quadriceps strength using a portable dynamometer in kilogram-force (kgf)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Figueiredo Alves da Silva, PT, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No